CLINICAL TRIAL: NCT03853798
Title: An Open-Label, Multicenter, Extension Study of AG-348 in Adult Subjects With Pyruvate Kinase Deficiency Previously Enrolled in AG-348 Studies
Brief Title: Extension Study of AG-348 in Adult Participants With Pyruvate Kinase Deficiency Previously Enrolled in AG-348-006 or AG348-C-007
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG348-C-011; 2018-003459-39 (EudraCT Number)
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Pyruvate Kinase Deficiency
MeSH Terms: conditions — Pyruvate Kinase Deficiency of Red Cells | interventions — mitapivat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants who received placebo in Study AG348-C-006 and met the eligibility criteria of this extension study were enrolled to receive mitapivat tablets, 5 milligrams (mg), twice daily (BID), administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined at Week 12, and participants then received that optimized dose for a period of 12 weeks (Weeks 13-24) as a fixed dose and from Week 25 to Week 193, until study withdrawal, or the study was closed.
  Interventions: Drug: Mitapivat
- Cohort 2 (Experimental): Participants who received mitapivat at a dose of 5 mg, 20 mg, or 50 mg, BID, in the fixed dose period of Study AG348-C-006 and met the eligibility criteria of this extension study continued to receive the same mitapivat dose up to Week 193 or until study withdrawal, or the study was closed.
  Interventions: Drug: Mitapivat
- Cohort 3 (Experimental): Participants who received mitapivat at a dose of 5 mg, 20 mg, or 50 mg, BID, in the fixed dose period of Study AG348-C-007 and met the eligibility criteria of this extension study continued to receive the same mitapivat dose up to Week 193 or until study withdrawal, or the study was closed.
  Interventions: Drug: Mitapivat

INTERVENTIONS:
Drug: Mitapivat — Tablets
  Other Names: AG-348; AG-348 sulfate hydrate; Mitapivat sulfate

SUMMARY:
This is an open-label, multicenter, extension study to evaluate the long-term safety, tolerability, and efficacy of treatment with mitapivat in participants who were previously enrolled in Study AG348-C-006 or Study AG348-C-007.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to comply with study visits and procedures.
* Have signed written informed consent prior to participating in this extension study.
* Have completed either antecedent study AG348-C-006 or AG348-C-007 through the Part 2 Week 24 Visit.
* Cohorts 2 and 3: Have demonstrated clinical benefit from mitapivat treatment in the antecedent study, in the opinion of the Investigator.
* For women of reproductive potential, have a negative pregnancy test during screening of this extension study.
* For women of reproductive potential as well as men with partners who are women of reproductive potential, be abstinent as part of their usual lifestyle, or agree to use 2 forms of contraception, 1 of which must be considered highly effective, from the time of giving informed consent, during the study, and for 28 days following the last dose of study drug for women and 90 days following the last dose of study drug for men.

Exclusion Criteria:

* Have a significant medical condition (including clinically significant laboratory abnormality) that developed during his/her antecedent AG- 348 study that confers an unacceptable risk to participating in this extension study, that could confound the interpretation of the study data, and/or that compromises the ability of the participant to complete study visits and procedures.
* Are currently pregnant or breastfeeding.
* Have a splenectomy scheduled during the study treatment period.
* Meet the withdrawal criteria of his/her antecedent mitapivat study during screening of this extension study.
* Are currently receiving medications that are strong inhibitors of cytochrome P450 (CYP)3A4 that have not been stopped for a duration of at least 5 days or a time frame equivalent to 5 half-lives (whichever is longer) before start of study drug; or strong inducers of CYP3A4 that have not been stopped for a duration of at least 28 days or a time frame equivalent to 5 half-lives (whichever is longer) before start of study drug on this extension study.
* Have received anabolic steroids, including testosterone preparations, within 28 days prior to start of study drug on this extension study.
* Have received hematopoietic stimulating agents (eg, erythropoietins, granulocyte colony stimulating factors, thrombopoietins) within 28 days prior to start of study drug on this extension study.
* Have exposure to any investigational drug other than mitapivat, device, or procedure within 3 months prior to start of study drug on this extension study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (42):
- United States (12):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - UCSF Benioff Children's Hospital, Oakland, Oakland, California
  - Emory-Children's Center, Atlanta, Georgia
  - Indiana Hemophilia & Thrombosis Center Inc., Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Wayne State University School of Medicine, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Houston Methodist Research Institute, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
- UNICAMP - Hemocentro, São Paulo, Brazil
- McMaster University, Hamilton, Ontario, Canada
- Herlev University Hospital, Herlev, Denmark
- France (4):
  - CHU Hopitaux de Bordeaux - Hôpital Saint-André, Bordeaux
  - CHU Hôpital Henri Mondor, Créteil
  - Hospital La Timone, Marseille
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
- Germany (2):
  - Charite - UB - CVK - Medizinische Klinik, Berlin
  - Universitätsklinik Würzburg, Würzburg
- St James's Hospital, Dublin, Ireland
- Italy (4):
  - Ospedale Galliera, Genova
  - Osp Maggiore Policlinico Milano, Milan
  - AORN Cardarelli, Napoli
  - Università della Campania "Luigi Vanvitelli", Napoli
- Japan (5):
  - Mie University Hospital, Tsu, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Kyoto Katsura Hospital, Kyoto
  - Kansai Medical University, Dep. of Pediatrics, Hirakata Hospital, Osaka
  - Toho University Omori Medical Center, Tokyo
- Van Creveldkliniek, Utrecht, Netherlands
- Yeungnam University Hospital, Daegu, South Korea
- Spain (3):
  - Hospital. U. Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Htal Clínico Universitario Virgen de la Arrixaca., Murcia
- Centre Hospitalier Universitaire Vaudois (CHUV), Vaud (Lausanne), Switzerland
- Faculty of Medicine Siriraj Hospital, Bangkok, Thailand
- Hacettepe University Faculty of Medicine, Ankara, Turkey (Türkiye)
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge
  - Imperial College Healthcare NHS Trust, London
  - University College London, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Beers EJ, Al-Samkari H, Grace RF, Barcellini W, Glenthoj A, DiBacco M, Wind-Rotolo M, Xu R, Beynon V, Patel P, Porter JB, Kuo KHM. Mitapivat improves ineffective erythropoiesis and iron overload in adult patients with pyruvate kinase deficiency. Blood Adv. 2024 May 28;8(10):2433-2441. doi: 10.1182/bloodadvances.2023011743. PMID 38330179
- [Derived] Rab MAE, Van Oirschot BA, Kosinski PA, Hixon J, Johnson K, Chubukov V, Dang L, Pasterkamp G, Van Straaten S, Van Solinge WW, Van Beers EJ, Kung C, Van Wijk R. AG-348 (Mitapivat), an allosteric activator of red blood cell pyruvate kinase, increases enzymatic activity, protein stability, and ATP levels over a broad range of PKLR genotypes. Haematologica. 2021 Jan 1;106(1):238-249. doi: 10.3324/haematol.2019.238865. PMID 31974203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 42 investigative sites in Denmark, France, Italy, Spain, Germany, United Kingdom, Netherlands, Ireland, Switzerland, United States, Canada, Japan, Korea, Thailand, Brazil and Turkey from 21 March 2019 to 03 July 2024.
Pre-assignment Details: A total of 90 participants who had completed Study AG348-C-006 (NCT03548220) or AG348-C-007 (NCT03559699), were enrolled in this extension study to receive mitapivat treatment. Participants were assigned to Cohorts 1, 2 or 3 depending on the previous treatment received in the antecedent studies.
Groups:
- Cohort 1: 5 mg: Participants who received placebo in Study AG348-C-006 and met the eligibility criteria of this extension study were enrolled to receive mitapivat tablets, 5 milligrams (mg), twice daily (BID), administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined as 5 mg, BID, at Week 12, which was followed for a period of 12 weeks (Weeks 13-24) as a fixed dose and then from Week 25 to Week 193, until study withdrawal, or the study was closed.
- Cohort 1: 20 mg: Participants who received placebo in Study AG348-C-006 and met the eligibility criteria of this extension study were enrolled to receive mitapivat tablets, 5 mg, BID, administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined as 20 mg, BID, at Week 12, which was followed for a period of 12 weeks (Weeks 13-24) as a fixed dose and then from Week 25 to Week 193, until study withdrawal, or the study was closed.
- Cohort 1: 50 mg: Participants who received placebo in Study AG348-C-006 and met the eligibility criteria of this extension study were enrolled to receive mitapivat tablets, 5 mg, BID, administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined as 50 mg, BID, at Week 12, which was followed for a period of 12 weeks (Weeks 13-24) as a fixed dose and then from Week 25 to Week 193, until study withdrawal, or the study was closed.
- Cohort 2: 5 mg: Participants who received mitapivat at a dose of 5 mg, BID, in the fixed dose period of Study AG348-C-006 and met the eligibility criteria of this extension study continued to receive the same mitapivat dose up to Week 193 or until study withdrawal, or the study was closed.
- Cohort 2: 20 mg: Participants who received mitapivat at a dose of 20 mg, BID, in the fixed dose period of Study AG348-C-006 and met the eligibility criteria of this extension study continued to receive the same mitapivat dose up to Week 193 or until study withdrawal, or the study was closed.
- Cohort 2: 50 mg: Participants who received mitapivat at a dose of 50 mg, BID, in the fixed dose period of Study AG348-C-006 and met the eligibility criteria of this extension study continued to receive the same mitapivat dose up to Week 193 or until study withdrawal, or the study was closed.
- Cohort 3: 5 mg: Participants who received mitapivat at a dose of 5 mg, BID, in the fixed dose period of Study AG348-C-007 and met the eligibility criteria of this extension study continued to receive the same mitapivat dose up to Week 193 or until study withdrawal, or the study was closed.
- Cohort 3: 20 mg: Participants who received mitapivat at a dose of 20 mg, BID, in the fixed dose period of Study AG348-C-007 and met the eligibility criteria of this extension study continued to receive the same mitapivat dose up to Week 193 or until study withdrawal, or the study was closed.
- Cohort 3: 50 mg: Participants who received mitapivat at a dose of 50 mg, BID, in the fixed dose period of Study AG348-C-007 and met the eligibility criteria of this extension study continued to receive the same mitapivat dose up to Week 193 or until study withdrawal, or the study was closed.
Period: Overall Study
Arm/Group | Cohort 1: 5 mg | Cohort 1: 20 mg | Cohort 1: 50 mg | Cohort 2: 5 mg | Cohort 2: 20 mg | Cohort 2: 50 mg | Cohort 3: 5 mg | Cohort 3: 20 mg | Cohort 3: 50 mg
Started | 1 | 1 | 36 | 2 | 3 | 30 | 0 | 1 | 16
Completed | 0 | 0 | 25 | 2 | 3 | 22 | 0 | 1 | 10
Not Completed | 1 | 1 | 11 | 0 | 0 | 8 | 0 | 0 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 4 | 0 | 0 | 5 | 0 | 0 | 4
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Approved Drug Available for Indication | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other un-specified | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of study treatment. Due to limited number of participants with optimal dose of 5 mg or 20 mg in antecedent studies AG348-C-006 (NCT03548220) and AG348-C-007 (NCT03559699), it was pre-specified in the statistical analysis plan (SAP) to report data for baseline characteristics by Cohort.
Groups:
- Cohort 1: Participants who received placebo in Study AG348-C-006 and met the eligibility criteria of this extension study were enrolled to receive mitapivat tablets, 5 mg, BID, administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined at Week 12, and participants then received that optimized dose for a period of 12 weeks (Weeks 13-24) as a fixed dose and from Week 25 to Week 193, until study withdrawal, or the study was closed.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 38 | 35 | 17 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.0 (15.95) | 36.9 (15.77) | 36.9 (15.09) | 37.4 (15.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 12 | 55
  Male | 15 | 15 | 5 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 33 | 23 | 12 | 68
  Unknown or Not Reported | 4 | 10 | 5 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31 | 23 | 13 | 67
  Asian | 3 | 5 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Other | 1 | 0 | 0 | 1
  Not reported | 3 | 6 | 2 | 11
Femoral Total: T-score [Mean (Standard Deviation); unit: T-score] — The T-score is the number of standard deviations that bone density is above or below the average. A score of greater than or equal to (≥) -1 indicates normal bone density, a score less than (<) -1 and greater than (>) -2.5 indicates a sign of osteopenia (bone density below normal), and a score less than or equal to (≤) -2.5 indicates a sign of osteoporosis. The baseline is the last assessment before start of study treatment (mitapivat). Population: Number analyzed is the number of participants that were evaluable for analysis at the baseline.
  T-score
    number analyzed (Participants) | 38 | 34 | 17 | 89
    (all) | -0.834 (1.1182) | -1.139 (1.0995) | -0.813 (0.6748) | -0.946 (1.0416)
Femoral Total: Z-score [Mean (Standard Deviation); unit: Z-score] — The Z-score is a statistical measure to describe whether a value was above or below the standard. A Z-score of 0 is equal to the standard. Lower numbers indicate values lower than the standard and higher numbers indicate values higher than the standard. The baseline is the last assessment before start of study treatment (mitapivat). Population: Number analyzed is the number of participants that were evaluable for analysis at the baseline.
  Z-score
    number analyzed (Participants) | 38 | 34 | 17 | 89
    (all) | -0.548 (1.1574) | -0.916 (1.0657) | -0.529 (0.7137) | -0.685 (1.0560)
Adjusted Spine: T-Score [Mean (Standard Deviation); unit: T-score] — The T-score is the number of standard deviations that bone density is above or below the average. A score of ≥ -1 indicates normal bone density; score between < -1 and > -2.5 indicates a sign of osteopenia (bone density below normal), and score of ≤ -2.5 indicates a sign of osteoporosis. The baseline is the last assessment before start of study treatment (mitapivat). Population: Number analyzed is the number of participants that were evaluable for analysis at the baseline.
  T-score
    number analyzed (Participants) | 38 | 34 | 17 | 89
    (all) | -1.143 (1.0926) | -1.808 (1.1589) | -1.161 (1.0469) | -1.400 (1.1440)
Adjusted Spine: Z-score [Mean (Standard Deviation); unit: Z-score] — The Z-score is a statistical measure to describe whether a value was above or below the standard. A Z-score of 0 is equal to the standard. Lower numbers indicate values lower than the standard and higher numbers indicate values higher than the standard. The baseline is the last assessment before start of study treatment (mitapivat). Population: Number analyzed is the number of participants that were evaluable for analysis at the baseline.
  Z-score
    number analyzed (Participants) | 38 | 34 | 17 | 89
    (all) | -0.804 (1.2529) | -1.536 (1.2469) | -0.848 (1.0420) | -1.092 (1.2506)

OUTCOME MEASURES:

1. Primary Outcome: All Cohorts: Number of Participants With at Least One Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, Related TEAEs and TEAEs With Severity Greater Than or Equal to Grade 3
Description: A clinical adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the study drug. TEAEs are AEs with an initial onset date during the on-treatment period or worsening from baseline and include both serious and non-serious TEAEs. Severity of AEs was evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE; Version 4.03): grade 1: mild; grade 2: moderate; grade 3: severe or medically significant but not immediately life-threatening; grade 4: life threatening or disabling; grade 5: death related to AE.
Time Frame: Up to 197 weeks
Population: The safety analysis set included all participants who received at least 1 dose of study treatment. Due to limited number of participants with optimal dose of 5 mg or 20 mg in antecedent studies AG348-C-006 (NCT03548220) and AG348-C-007 (NCT03559699), it was pre-specified in the SAP to report data for this outcome measure (OM) by Cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 38 | 35 | 17
Participants
  Participants with TEAEs | 37 | 33 | 15
  Participants with Serious TEAEs | 11 | 8 | 4
  Participants with TEAEs related to study drug | 22 | 14 | 4
  Participants with any TEAE of Grade ≥ 3 | 16 | 10 | 5

2. Primary Outcome: All Cohorts: Number of Participants With TEAEs Leading to Dose Reduction, Treatment Interruption and Treatment Discontinuation
Description: A clinical AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the study drug. TEAEs are AEs with an initial onset date during the on-treatment period or worsening from baseline and include both serious and non-serious TEAEs. Number of participants with TEAEs leading to dose reduction, treatment interruption and treatment discontinuation are reported.
Time Frame: Up to 197 weeks
Population: The safety analysis set included all participants who received at least 1 dose of study treatment. Due to limited number of participants with optimal dose of 5 mg or 20 mg in antecedent studies AG348-C-006 (NCT03548220) and AG348-C-007 (NCT03559699), it was pre-specified in the SAP to report data for this OM by Cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 38 | 35 | 17
Participants
  Participants with TEAEs Leading to Dose Reduction | 2 | 2 | 1
  Participants with TEAEs Leading to Interruption | 3 | 4 | 0
  Participants with TEAEs Leading to Discontinuation | 2 | 1 | 0

3. Primary Outcome: All Cohorts: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters Reported as Grade Greater Than or Equal to (≥)3 TEAEs
Description: Clinical laboratory assessments including hematology, clinical chemistry, triglycerides, urate, coagulation, urinalysis, and liver function tests were performed in the study. Clinically significant treatment-emergent laboratory abnormalities were graded according to the NCI CTCAE; Version 4.03: grade 1: mild; grade 2: moderate; grade 3: severe or medically significant but not immediately life-threatening; grade 4: life threatening or disabling; grade 5: death related to AE. Clinical significance was determined based on the judgment of the Investigator.
Time Frame: Up to 197 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 38 | 35 | 17
Participants
  Anaemia | 3 | 1 | 0
  Haemolysis | 1 | 2 | 0
  Alanine aminotransferase increased | 0 | 0 | 1
  Aspartate aminotransferase increased | 2 | 1 | 1
  Blood bilirubin increased | 0 | 0 | 1
  Blood triglycerides increased | 1 | 0 | 0
  Hypertriglyceridaemia | 1 | 0 | 0

4. Primary Outcome: All Cohorts: Number of Participants With Clinically Significant Abnormalities in Vital Signs Measurements and Physical Examinations Reported as TEAEs
Description: Vital signs and physical examinations including height, weight, body mass index (BMI), systolic blood pressure, diastolic blood pressure, pulse rate, temperature were assessed. Number of participants who experienced clinically significant abnormalities in vital signs and physical examinations as TEAEs were reported. Clinical significance was determined based on the judgment of the Investigator.
Time Frame: Up to 197 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 38 | 35 | 17
Participants
  Weight decreased | 0 | 1 | 1
  Hot flush | 2 | 0 | 2
  Hypotension | 1 | 0 | 0
  Hypertension | 1 | 2 | 0

5. Primary Outcome: All Cohorts: Number of Participants With Clinically Significant Abnormalities in Bone Mineral Density (BMD)
Description: BMD was measured by dual-energy X-ray absorptiometry (DXA) scans during the study. Number of participants with clinically significant abnormalities were reported. Clinical significance was determined based on the judgment of the Investigator.
Time Frame: Up to 192 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 38 | 35 | 17
Participants | 0 | 1 | 0

6. Primary Outcome: All Cohorts: Change From Baseline in Adjusted Spine T-score
Description: T-score of adjusted spine were assessed by DXA scans. The T-score is the number of standard deviations that bone density is above or below the average. A score of ≥ -1 indicates normal bone density; score between < -1 and > -2.5 indicates a sign of osteopenia (bone density below normal), and score of ≤ -2.5 indicates a sign of osteoporosis.
Time Frame: Baseline, Week 192
Population: The safety analysis set included all participants who received at least 1 dose of study treatment. Here, overall number of participants analyzed indicates the number of participants who were evaluable for this OM. Due to limited number of participants with optimal dose of 5 mg or 20 mg in antecedent studies AG348-C-006 (NCT03548220) and AG348-C-007 (NCT03559699), it was pre-specified in the SAP to report data for this OM by Cohort.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 24 | 20 | 8
T-score | 0.046 (0.4874) | 0.234 (0.4383) | 0.416 (1.1090)

7. Primary Outcome: All Cohorts: Change From Baseline in Adjusted Spine Z-score
Description: The Z-score is a statistical measure to describe whether a value was above or below the standard. A Z-score of 0 is equal to the standard. Lower numbers indicate values lower than the standard and higher numbers indicate values higher than the standard.
Time Frame: Baseline, Week 192
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 24 | 20 | 8
Z-score | 0.152 (0.4585) | 0.332 (0.4002) | 0.530 (1.2409)

8. Primary Outcome: All Cohorts: Change From Baseline in Femoral Total T-score
Description: T-score of femoral total were assessed by DXA scans. The T-score is the number of standard deviations that bone density is above or below the average. A score of ≥ -1 indicates normal bone density; score between < -1 and > -2.5 indicates a sign of osteopenia (bone density below normal), and score of ≤ -2.5 indicates a sign of osteoporosis.
Time Frame: Baseline, Week 192
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 24 | 20 | 8
T-score | -0.020 (0.2612) | 0.047 (0.3893) | 0.114 (0.5050)

9. Primary Outcome: All Cohorts: Change From Baseline in Femoral Total Z-score
Description: as for outcome 7
Time Frame: Baseline, Week 192
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Z- score
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 24 | 20 | 8
Z- score | 0.054 (0.2468) | 0.126 (0.3631) | 0.214 (0.5099)

10. Primary Outcome: All Cohorts: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG) Parameters Reported as TEAEs
Description: The following ECG parameters including RR, PR, heart rate-corrected QT interval using the Fridericia's formula (QRS), QT, and QTc were assessed during the study. Number of Participants with clinically significant abnormalities in ECG parameters as TEAEs were reported. Clinical significance was determined based on the judgment of the Investigator.
Time Frame: Up to 197 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 38 | 35 | 17
Participants | 0 | 1 | 0

11. Secondary Outcome: Cohort 1: Percentage of Participants Who Achieved a Hemoglobin (Hb) Response
Description: The Hb response was defined as a greater than or equal to (≥)1.5 grams per deciliter (g/dL) (0.93 millimoles per liter [mmol/L]) increase in Hb concentration from baseline that is sustained at 2 or more scheduled assessments, excluding those within 2 months (61 days) of transfusion. The baseline value for cohort 1 participants was the average of all available measurements from the central laboratory within 45 (42+3) days before start of study treatment in study AG348-C-011, excluding values within 61 days after a transfusion, or the baseline value from study AG348-C-006 if no assessment is available.
Time Frame: Baseline up to Week 24
Population: FAS included all participants who received at least 1 dose of study treatment. Due to limited number of participants with optimal dose of 5 mg or 20 mg in antecedent Study AG348-C-006 (NCT03548220), it was pre-specified in the SAP to report data for this OM by Cohort. As per planned analysis, data for this OM was reported for Cohort 1 only based on FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 38
percentage of participants | 39.5

12. Secondary Outcome: Cohort 1: Average Change From Baseline in Hb Concentration at Weeks 16, 20, and 24
Description: The baseline value for participants was the average of all available measurements from the central laboratory within 45 (42+3) days before start of study treatment in study AG348-C-011, excluding values within 61 days after a transfusion, or the baseline value from study AG348-C-006 if no assessment is available. The mean of average change from baseline in Hb concentration across Weeks 16, 20 and 24 is reported.
Time Frame: Baseline, Weeks 16, 20, and 24
Population: FAS included all participants who received at least 1 dose of study treatment. Overall number of participants analyzed indicates number of participants were evaluable for this OM. Due to limited number of participants with optimal dose of 5 mg or 20 mg in antecedent study AG348-C-006 (NCT03548220), it was pre-specified in the SAP to report data for this OM by Cohort. As per planned analysis, data for this OM was reported for Cohort 1 only based on FAS.
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Cohort 1
Number analyzed (Participants) | 36
grams per liter | 16.45 (15.634)

13. Secondary Outcome: Cohort 1: Area Under the Plasma Concentration-Time Curve From Time Zero to 8-hours Post-dose (AUC0-8) of Mitapivat
Time Frame: Pre-dose, 0.5, 1, 2, 4, and 8 hours post-dose at Week 12
Population: PK analysis population: all participants who were enrolled & received at least 1 dose of mitapivat with at least 1 nonzero plasma concentration of mitapivat at Week 12 visit. Overall number of participants analyzed: number of participants who received 50 mg BID mitapivat in Cohort 1 and were evaluable for this OM. As per planned analysis, data for this OM was reported by cohort and for Cohort 1 only based on FAS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms per milliliter (hr*ng/mL)
Arm/Group | Cohort 1
Number analyzed (Participants) | 23
hour*nanograms per milliliter (hr*ng/mL) | 3016 (27.5)

14. Secondary Outcome: Cohort 1: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC0-last) of Mitapivat
Time Frame: Pre-dose, 0.5, 1, 2, 4, and 8 hours post-dose at Week 12
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Cohort 1
Number analyzed (Participants) | 28
hr*ng/mL | 2990 (26.3)

15. Secondary Outcome: Cohort 1: Maximum Observed Plasma Concentration (Cmax) of Mitapivat
Time Frame: Pre-dose, 0.5, 1, 2, 4, and 8 hours post-dose at Week 12
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Cohort 1
Number analyzed (Participants) | 30
nanograms/milliliter (ng/mL) | 1018 (22.5)

16. Secondary Outcome: Cohort 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Mitapivat
Time Frame: Pre-dose, 0.5, 1, 2, 4, and 8 hours post-dose at Week 12
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1
Number analyzed (Participants) | 30
hours | 1.00 [0.45 to 4.3]

17. Secondary Outcome: Cohort 1: Time of Last Quantifiable Concentration (Tlast) of Mitapivat
Time Frame: Pre-dose, 0.5, 1, 2, 4, and 8 hours post-dose at Week 12
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1
Number analyzed (Participants) | 28
hours | 7.61 [3.57 to 8.53]

18. Secondary Outcome: Cohort 1: Plasma Concentration (Ctrough) at the End of a Dosing Interval of Mitapivat
Time Frame: Pre-dose, 0.5, 1, 2, 4, and 8 hours post-dose at Week 12
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1
Number analyzed (Participants) | 28
ng/mL | 62.8 (72.7)

19. Secondary Outcome: Cohort 1: Exposure-response (E-R) Relationship Between Safety Parameters and Mitapivat Concentration and Relevant Mitapivat Pharmacokinetic Parameters
Time Frame: First dose to up to 24 weeks
Population: After the dose optimization period, the 5 mg and 20 mg doses each had a single participant and the 50 mg dose had 36 participants. The exposure-relationship analysis planned cannot be performed with a single participant in multiple groups.
Measure: Mean (95% Confidence Interval); unit: Percent probability
Arm/Group | Cohort 1: 5 mg | Cohort 1: 20 mg | Cohort 1: 50 mg
Number analyzed (Participants) | 1 | 1 | 36
Percent probability | NA [NA to NA] — After the dose optimization period, the 5 mg and 20 mg doses each had a single participant and the 50 mg dose had 36 participants. The exposure-relationship analysis planned cannot be performed with a single participant in multiple groups. | NA [NA to NA] — After the dose optimization period, the 5 mg and 20 mg doses each had a single participant and the 50 mg dose had 36 participants. The exposure-relationship analysis planned cannot be performed with a single participant in multiple groups. | NA [NA to NA] — After the dose optimization period, the 5 mg and 20 mg doses each had a single participant and the 50 mg dose had 36 participants. The exposure-relationship analysis planned cannot be performed with a single participant in multiple groups.

20. Secondary Outcome: Cohorts 1 and 2: Change From Baseline in Hb Concentration
Description: The baseline value for cohort 1 participant was the average of all available measurements from the central laboratory within 45 (42+3) days before start of study treatment in study AG348-C-011, excluding values within 61 days after a transfusion, or the baseline value from study AG348-C-006 if no assessment was available. The baseline value for cohort 2 was from Study AG348-C-006.
Time Frame: Baseline, Week 192
Population: FAS included all participants who received at least 1 dose of study treatment. Here, overall number of participants analyzed indicates the number of participants who were evaluable for this OM. Due to limited number of participants with optimal dose of 5 mg or 20 mg in antecedent study AG348-C-006 (NCT03548220), it was pre-specified in the SAP to report data for this OM by Cohort. As per planned analysis, data for this OM was reported for Cohort 1 and 2 only based on FAS.
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 23
grams per liter | 22.39 (21.211) | 21.32 (20.721)

21. Secondary Outcome: Cohorts 1 and 2: Change From Baseline in Indirect Bilirubin
Description: The baseline value for cohort 1 participant was the average of all available measurements from the central laboratory within 45 (42+3) days before start of study treatment in study AG348-C-011, excluding values within 61 days after a transfusion, or the baseline value from study AG348-C-006 if no assessment is available. The baseline value for cohort 2 was from Study AG348-C-006.
Time Frame: Baseline, Week 192
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: micromoles per liter (μmol/L)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 21
micromoles per liter (μmol/L) | -57.50 (54.542) | -36.73 (35.511)

22. Secondary Outcome: Cohorts 1 and 2: Change From Baseline in Lactate Dehydrogenase (LDH)
Description: as for outcome 20
Time Frame: Baseline, Week 192
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Units per Liter (U/L)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 24 | 22
Units per Liter (U/L) | -46.10 (75.310) | -130.80 (275.424)

23. Secondary Outcome: Cohorts 1 and 2: Change From Baseline in Haptoglobin Levels
Description: as for outcome 20
Time Frame: Baseline, Week 192
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 24 | 25
grams per liter | 0.254 (0.4340) | 0.250 (0.4689)

24. Secondary Outcome: Cohorts 1 and 2: Change From Baseline in Reticulocytes/Erythrocytes Ratio
Description: The baseline value for Cohort 1 participants was the average of all available measurements from the central laboratory within 45 (42+3) days before start of study treatment in study AG348-C-011, excluding values within 61 days after a transfusion, or the baseline value from study AG348-C-006 if no assessment was available. The baseline value for Cohort 2 was from Study AG348-C-006.
Time Frame: Baseline, Week 192
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Reticulocytes/Erythrocytes Ratio
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 20
Reticulocytes/Erythrocytes Ratio | -0.1696 (0.16243) | -0.1565 (0.14631)

25. Secondary Outcome: Cohort 3: Change From Baseline in Number of Transfusion Episodes
Description: Number of transfusions at baseline was determined based on the transfusion data during the 52 weeks before informed consent for Cohort 3. Number of on-study transfusions was based on transfusions collected up to the end of the fixed dose period and standardized to 52 weeks. The change from baseline in number of transfusions was summarized for Cohort 3.
Time Frame: Baseline, Week 192
Population: FAS included all participants who received at least 1 dose of study treatment. Due to limited number of participants with optimal dose of 5 mg or 20 mg in antecedent study AG348-C-007 (NCT03559699), it was pre-specified in the SAP to report data for this OM by Cohort. As per planned analysis, data for this OM was reported for Cohort 3 only based on FAS.
Measure: Mean (Standard Deviation); unit: number of transfusion episodes
Arm/Group | Cohort 3
Number analyzed (Participants) | 17
number of transfusion episodes | 4.14 (5.487)

26. Secondary Outcome: Cohort 3: Change From Baseline in Number of Red Blood Cell (RBC) Units Transfused
Description: Annualized total number of RBC units transfused (units/52-week) during the study, including data up to end of study (EOS), was the total number of RBC units transfused during the entire study*52 / [(date of EOS - date of start of study treatment + 1)/7]. Number of RBC units were determined based on the transfusion data during the 52 weeks before informed consent of the antecedent study for Cohort 3. Number of on-study RBC units was based on transfusion data collected up to the end of the fixed dose period and standardized to 52 weeks.
Time Frame: Baseline, Week 192
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: number of RBC units transfused
Arm/Group | Cohort 3
Number analyzed (Participants) | 17
number of RBC units transfused | 7.25 (7.915)

27. Secondary Outcome: All Cohorts: Change From Baseline in Health-Related Quality of Life (HRQoL) Patient-Reported Outcome (PRO) Scores: Pyruvate Kinase Deficiency Diary (PKDD)
Description: The PKDD is a validated, daily 7-item PRO instrument with a recall period of 24 hours that measures the core signs and symptoms associated with pyruvate kinase deficiency in adults. The symptoms include tiredness, jaundice, bone pain, shortness of breath, and energy level. PKDD daily scores were calculated based on the participant's response to the PKDD questionnaire. Score ranges from 25 to 76, with higher scores indicating more severe symptoms and a higher disease burden. The change from baseline in weekly mean scores was summarized. A negative change from baseline indicates a lower disease burden. Baseline of weekly mean score was defined as average of daily scores collected within 7 days before start of study treatment (mitapivat). For Cohort 1, last measurement before the start of study treatment in AG348-C-011 was used as baseline; if baseline was missing, then baseline value from AG348-C-006 was used. For Cohorts 2 & 3 baseline values from -006 and-007, respectively, were used.
Time Frame: Baseline, Week 24
Population: FAS included all participants who received at least 1 dose of study treatment. Here, overall number of participants analyzed indicates the number of participants who were evaluable for this OM. Due to limited number of participants with optimal dose of 5 mg or 20 mg in antecedent studies AG348-C-006 (NCT03548220) and AG348-C-007 (NCT03559699), it was pre-specified in the SAP to report data for this OM by Cohort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 24 | 10
score on a scale | -3.75 (5.805) | -6.09 (7.617) | -5.04 (12.273)

28. Secondary Outcome: All Cohorts: Change From Baseline in HRQoL PRO Scores: Pyruvate Kinase Deficiency Impact Assessment (PKDIA)
Description: PKDIA is a 12-item PRO measure of common impacts of PK deficiency on activities of daily living. Participants rated how PK deficiency has impacted aspects of daily living in past 7 days, including impacts on relationships & leisure and social, mental, and physical activities. PKDIA score at each visit was based on 8 items that were retained after in-trial psychometric validation and calculated at each visit based on participant's response to PKDIA questionnaire. Score ranges from 30 to 76, with higher scores indicating higher disease burden. Negative change from baseline indicates lower disease burden. Baseline was defined as the last complete assessment (with no missing item in response) before start of study treatment. For Cohort 1, last measurement before start of study treatment in AG348-C-011 was used as baseline; if baseline was missing, then baseline value from AG348-C-006 was used. For Cohorts 2 and 3, the baseline values from 006 and 007, respectively, were used.
Time Frame: Baseline, Week 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 31 | 28 | 14
score on a scale | -3.9 (7.38) | -6.6 (8.75) | -5.4 (12.83)

ADVERSE EVENTS:
Time Frame: Up to 197 weeks
Description: The safety analysis set included all participants who received at least 1 dose of study treatment.
Groups:
- Cohort 1: 5 mg: Participants who received placebo in Study AG348-C-006 and met the eligibility criteria of this extension study were enrolled to receive mitapivat tablets, 5 mg, BID, administered orally, for 4 weeks as a starting dose, followed by two potential sequential dose level increases to 20 mg and 50 mg BID at Weeks 4 and 8 respectively as determined by the investigator based on safety and efficacy. The optimized dose for each participant was determined as 5 mg, BID, at Week 12, which was followed for a period of 12 weeks (Weeks 13-24) as a fixed dose and then from Week 25 to Week 193, until study withdrawal, or the study was closed.
Arm/Group | Cohort 1: 5 mg | Cohort 1: 20 mg | Cohort 1: 50 mg | Cohort 2: 5 mg | Cohort 2: 20 mg | Cohort 2: 50 mg | Cohort 3: 5 mg | Cohort 3: 20 mg | Cohort 3: 50 mg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/36 | 0/2 | 0/3 | 1/30 | 0/0 | 0/1 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 10/36 | 0/2 | 2/3 | 6/30 | 0/0 | 0/1 | 4/16
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 35/36 | 2/2 | 2/3 | 27/30 | 0/0 | 1/1 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 5 mg (N=1) | Cohort 1: 20 mg (N=1) | Cohort 1: 50 mg (N=36) | Cohort 2: 5 mg (N=2) | Cohort 2: 20 mg (N=3) | Cohort 2: 50 mg (N=30) | Cohort 3: 5 mg (N=0) | Cohort 3: 20 mg (N=1) | Cohort 3: 50 mg (N=16)
Sepsis (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vascular stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 5 mg (N=1) | Cohort 1: 20 mg (N=1) | Cohort 1: 50 mg (N=36) | Cohort 2: 5 mg (N=2) | Cohort 2: 20 mg (N=3) | Cohort 2: 50 mg (N=30) | Cohort 3: 5 mg (N=0) | Cohort 3: 20 mg (N=1) | Cohort 3: 50 mg (N=16)
COVID-19 (Infections and infestations) | 0 | 0 | 12 | 1 | 2 | 13 | 0 | 1 | 5
Nasopharyngitis (Infections and infestations) | 0 | 0 | 6 | 1 | 0 | 5 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 9 | 0 | 0 | 4 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 4
Influenza (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 3 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 3
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 3 | 0 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear lobe infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Helminthic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Implant site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infective tenosynovitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 10 | 1 | 1 | 6 | 0 | 0 | 4
Pyrexia (General disorders) | 0 | 0 | 10 | 2 | 0 | 7 | 0 | 0 | 3
Influenza like illness (General disorders) | 0 | 0 | 4 | 0 | 1 | 1 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 9 | 0 | 2 | 5 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 0 | 1 | 2 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 1 | 0 | 2 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 1 | 3 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 20 | 2 | 0 | 6 | 0 | 1 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 1
Anosmia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2
Migraine (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 6 | 0 | 1 | 4 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 6 | 0 | 0 | 3 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 1 | 4 | 0 | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 0 | 0 | 2 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 0 | 2 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 8 | 1 | 0 | 4 | 0 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 6 | 1 | 0 | 2 | 0 | 0 | 4
Vitamin D decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
High density lipoprotein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver iron concentration increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Middle insomnia (Psychiatric disorders) | 0 | 0 | 8 | 0 | 0 | 2 | 0 | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 3 | 0 | 1 | 3
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 1 | 2 | 0 | 0 | 1
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 1 | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipohaemarthrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 5 | 0 | 0 | 2 | 0 | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Perineal cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meibomian gland dysfunction (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The information obtained from the clinical study will be used towards the development of mitapivat and may be disclosed to regulatory authority(ies), other Investigators, corporate partners, or consultants as required.

DOCUMENTS (2):
  • Study Protocol (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT03853798/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT03853798/SAP_001.pdf